CLINICAL TRIAL: NCT06854861
Title: Premixed Glucagon/Insulin Solution for Faster Insulin Absorption in Type 1 Diabetes
Acronym: MicroGlucag2
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No sign of anticipated effect.
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MicroGlucagon2; 2023-510408-32-02 (EU CTIS Number)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: One day with Lyumjev and one day with premixed Lyumjev in each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyumjev (Active Comparator): Lyumjev 0.1 Unit /kg body weight
  Interventions: Drug: Lyumjev 100 UNT/ML Injectable Solution
- Premixed Lyumjev (Experimental): Lyumjev 0.1 Unit /kg body weight. Lyumjev is premixed with 5 ng glucagon/Unit insulin
  Interventions: Drug: Premixed Lyumjev

INTERVENTIONS:
Drug: Lyumjev 100 UNT/ML Injectable Solution — 0.1 unit insulin Lyumjev /kg body weight is injected subcutaneously
  Other Names: Lyumjev
  Arms: Lyumjev
Drug: Premixed Lyumjev — A solution of 5 ng glucagon /Unit Lyumjev is injcetd subcutaneously. 0.1 unit insulin / kg body weight is used.
  Arms: Premixed Lyumjev

SUMMARY:
We will investigate if Lyumjev premixed with nanogram amounts of glucagon speed up the absorption of insulin and the effect on whole body glucose consumption compared to native lyumjev in patients with type 1 diabetes. To do that we will perform euglycemic clamps investigations in patients meetinng fasting in the morning on two separate days.Frequent samples for glucose and insulin measuremenst will be drawn and the day with lyumjev only will be compared to the day with premixed Lyumjev.

DETAILED DESCRIPTION:
Rationale:

We recently published that in healthy subjects, micro-doses of glucagon significantly increase local subcutaneous (SC) blood flow. As the absorption of insulin among other factors also depend on the local subcutaneous blood flow, we hypothesised that micro-doses of glucagon at the site of SC insulin delivery enhance the absorption of insulin and speed up the effect on blood glucose levels. Recently, in anesthetized pigs we found that adding 0.1 mg of glucagon at the site of SC insulin injection enhances the insulin absorption and we have unpublished animal data confirming that micro-doses of glucagon premixed in insulin (Lyumjev®) enhances the absorption of SC injected insulin. Thus, we hypothesize that adding micro-amounts of glucagon to an insulin solution will speed up the absorption of insulin and the effect on glucose metabolism.

Objective To study if adding micro-amounts of glucagon to a fast-acting insulin (Lyumjev®) before injection speed up the absorption of and effect on glucose metabolism of SC injected insulin.

Trial design Open, prospective, controlled, single centre investigation where patients with T1D are their own controls. They will meet fasting in the morning on two separate days and receive a SC injection with insulin on both days. One of the days they will be randomised to receive an insulin solution where 5 ng glucagon per unit insulin has been added.

Intervention Participants are asked to fast from midnight before entering the research facility at 08 in the morning. On the morning of the study days patients will be asked to adjust the insulin infusion to have a glucose around 6.0 mmol/L when arriving at the research facility. When arriving the pump will be shut down, and

1. If glucose is >6.0 mmol/L intravenous (IV) insulin will be given (guided by a physician) for up to 2 hour to stabilize glucose levels at 6.0 mmol/L.
2. If glucose is <6.0 mmol/L IV glucose is given for up to 2 hours to stabilize glucose levels at 6.0 mmol/L.

An indwelling intravenous catheter is established, and glucose is measured every 5 minutes for at least 20 minutes before the injection with study insulin or glucagon/insulin solution. Another intravenous access is also established and used for continuous glucose infusion (euglycemic clamp procedure).

The dose of insulin (Lyumjev®) or glucagon/insulin (glucagon/Lyumjev®) solution (5 ng glucagon/Unit insulin) will be 0.1 unit of insulin per kg body weight. The same dose of insulin is used on both study days.

ELIGIBILITY:
Inclusion Criteria:

1. T1D for at least one year.
2. Age 18 - 70 years.
3. Last known HbA1c <75 mmol/mol (< 9.0%).
4. Treated with an insulin pump or a hybrid artificial pancreas (AP).

Exclusion criteria:

1. Pregnant women or women trying to conceive (women will not be screened by a pregnancy test).
2. Any chronic disease, including psychiatric illnesses, judged incompatible with participation in the study.
3. Unfit for participation for any reason as judged by the investigators.
4. Known hypersensitivity to glucagon or to any of the excipients of the drug formulations.
5. Known phaeochromocytoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the glucose consumption curve | First 30 minutes
  Area under the glucose consumption curve
Area under the insulin curve Area under the insulin curve | First 30 minutes
  Area under the insulin curve

SECONDARY OUTCOMES:
Area under the glucose consumption curve | Any time frame from 0 to 4 hours
  Area under the glucose consumption curve
Area under the insulin curve | Any time frame from 0 to 4 hours
  Area under the insulin curve

CONTACTS AND LOCATIONS:
Overall Officials: Sven M Carlsen, MD PhD, Principal Investigator — St. Olav/NTNU
Locations (1):
- St. Olavs University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No